CLINICAL TRIAL: NCT02974075
Title: Safety and Efficacy of Salvage Lymph Node Dissection in Prostate Cancer Patients With Nodal Recurrence After Radical Prostatectomy With Curative Intent - a Prospective Single Center Phase I/II Study
Brief Title: Salvage Lymph Node Dissection in Prostate Cancer Patients With Recurrence After Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Bernhard Grubmüller, MD, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1460/2016
Record Dates: First submitted 2016-11-20; First posted 2016-11-28 (Estimated); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer Recurrent

ARMS (1):
- Salvage lymph node dissection (Experimental): Patients will undergo extended pelvic salvage lymph node dissection
  Interventions: Procedure: Salvage lymph node dissection

INTERVENTIONS:
Procedure: Salvage lymph node dissection — Open pelvic surgery to dissect pelvic lymph nodes. The landmarks for dissection are: 1. Inferior mesenteric artery 2. Ilioinguinal nerve 3. Inguinal ligament 4. Dorsal pelvic floor 5. Urinary bladder

SUMMARY:
Despite continuous technical improvements in urologic surgery, up to 40% of prostate cancer patients will develop biochemical recurrence after radical prostatectomy (RP), potentially because of micro metastasis at the time of the primary surgery.

With improved radiological modalities and nuclear medicine tracers like 68Ga-PSMA PET/CT, which allow the localization of the site of recurrence, there is increasing interest in metastasis directed therapies, such as salvage lymph node dissection.

The pelvic extended salvage lymph node dissection (sLND) is a promising option for treating prostate cancer patients with local recurrence after radical prostatectomy with curative intent. Several retrospective series has been published to determine the local value of sLND. Despite the first data seem to be feasible and promising, to date no prospective evaluation has been made. Thus sLND is still experimental according to the guidelines and is considered as an off label therapy.

This prospective single center phase I/II study was conducted to investigate the safety and early efficacy of salvage lymph node dissection in prostate cancer patients with local pelvic recurrence after radical prostatectomy (RP) with curative intention.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients with lymph node metastasis in pelvic imaging
* Status post radical prostatectomy with curative intent
* Ability for informed consent
* No sign for bone or visceral metastasis
* Male > 18 years
* ECOG performance status 0 or 1

Exclusion Criteria:

* Male < 18 years
* No ability for informed consent
* Sign for bone or visceral metastasis
* Deep venous thrombosis or pulmonary embolism within the last 6 months before study screening
* ECOG performance status 2 or more

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2024-11 (Actual)

PRIMARY OUTCOMES:
The rate of periperative complications within 90 days after surgery | 90 days
The Prostate specific antigen value after 6 weeks. | 6 weeks

SECONDARY OUTCOMES:
Change in Prostate Specific Antigen doubling time | 2 years
Time until development of castration resistance | 2 years
Time until development of distant metastasis | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shahrokh Francois Shariat, MD, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria